CLINICAL TRIAL: NCT05137899
Title: Neoadjuvant Combination of Atezolizumab/Bevacizumab Versus Neoadjuvant Radiation Therapy Prior to Hepatectomy in Hepatocellular Carcinoma with Portal Vein Tumour Thrombus (ADVANCE HCC) Hoffmann La Roche Protocol Number: ML42525
Brief Title: Neoadjuvant Combination of Atezolizumab/Bevacizumab Versus Neoadjuvant Radiation Therapy
Acronym: ADVANCE HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges, Hoffman La Roche strategic priority shift
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2021-ADVANCE HCC ML42545
Record Dates: First submitted 2021-11-10; First posted 2021-11-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumour Thrombosis
Keywords: Neoadjuvant Atezolizumab/Bevacizumab; Neoadjuvant Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Neoadjuvant Atezolizumab/Bevacizumab versus neoadjuvant SBRT in patients with biopsy proven solitary HCC with PVTT involving the portal vein branches.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Atezolizumab/Bevacizumab (Experimental): • Arm 1: neoadjuvant atezolizumab 1200 mg IV q3weeks x 4 cycles, and bevacizumab 15 mg/kg IV q3weeks x 4 cycles
  Interventions: Combination Product: Neoadjuvant
- Neoadjuvant SBRT (Experimental): • Arm 2: neoadjuvant stereotactic body radiation therapy (SBRT), target volume 30 40 Gy, in 6-8 Gy per day over five days, delivered every other day
  Interventions: Combination Product: Neoadjuvant

INTERVENTIONS:
Combination Product: Neoadjuvant — Neoadjuvant atezolizumab/bevacizumab or neoadjuvant SBRT prior to hepatectomy

SUMMARY:
A multicentre, parallel group, randomized controlled Phase II clinical trial evaluating neoadjuvant Atezolizumab/Bevacizumab versus neoadjuvant SBRT in patients with biopsy proven solitary HCC with PVTT involving the portal vein branches. Both arms are considered experimental, and as such, a Simon two-stage design will be initially used within both arms. Only if both arms are deemed of interest for further study will a comparison between arms, using a pick-the-winner design, be conducted. Following the completion of neoadjuvant therapy, study participants will undergo a CT scan or MRI to assess tumour response to neoadjuvant therapy. Hepatic resection will be performed for those participants who meet the surgical resection criteria.

DETAILED DESCRIPTION:
Surgical resection without adjuvant therapy is the standard of care for most patients with solitary hepatocellular carcinoma (HCC). The presence of portal vein tumour thrombus (PVTT) is associated with a poor prognosis, and as a result patients usually do not undergo surgery.1 One potential strategy to improve the outcome of patients with HCC and PVTT is to administer treatment to the tumour prior to surgery, i.e. "neoadjuvant" therapy. This strategy has been proven to be effective in other types of cancer, and results in tumour downstaging and potentially eliminates micro-metastatic disease In a recent randomized controlled trial (RCT) in patients with HCC and PVTT, the addition of radiation therapy (RT) to the tumour prior to hepatic surgery was compared with surgery alone.4 There was a statistically significant improvement in survival with RT. Systemic therapy with the tyrosine kinase inhibitor Sorafenib improved survival compared to placebo in patients with advanced HCC and PVTT.5 Another recent trial in patients with advanced HCC demonstrated improved survival with the combination of Atezolizumab, an immune checkpoint inhibitor (ICI), and Bevacizumab, an antibody to vascular endothelial growth factor compared to Sorafenib alone.6

Currently, there is no standard of care for the neoadjuvant treatment of solitary HCC. Radiotherapy has not been widely adopted despite recent evidence suggesting some benefit. It is conceivable that RT will downsize the tumour increasing the surgical resection rate and reducing the shedding of tumour cells. Stereotactic Body Radiation Therapy (SBRT) is a type of RT that provides high dose, focal radiation to tumours using highly precise imaging and treatment fields, with rapid dose fall-off thereby sparing normal tissue. Based on experience in other cancers, it would seem judicious that effective systemic therapy be considered for the neoadjuvant treatment of HCC to downsize the primary tumour and eradicate occult micro-metastases.2,3

We hypothesize that treating patients with HCC and PVTT with either 1) neoadjuvant systemic therapy, or 2) neoadjuvant SBRT may lead to improved hepatic resection rates. Complete hepatic resection is being considered as a surrogate for good long-term outcomes. The aim of our randomized Phase II trial is to select the treatment arm with the most favourable outcomes based on a trade-off between resection rate and toxicity for study in a future trial.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven solitary HCC without biliary invasion, or metastases,
2. PVTT involving the portal vein branches: Vp1-Vp3 (Japanese Classification for HCC with PVTT, see Appendix II),
3. <10 cm maximal diameter on CT or MRI,
4. Child-Pugh Class A (see Appendix III), within 14 days prior to randomization. (All parameters without transfusion within 3 months).
5. Age > 18 years.

Exclusion Criteria:

1. Abnormal laboratory parameters (within 14 days of randomization):

   1. Hemoglobin < 90 g/L
   2. Platelet count < 75 x 109/L without transfusion
   3. INR >1.25
   4. Serum creatinine > 1.5 x ULN
   5. Urine dipstick for proteinuria > 2 (unless a 24-hour urine collection demonstrates < 1.5 g of protein in 24 hours.
2. Previous therapy for HCC:

   1. Systemic therapy, surgery or radiation therapy,
   2. Local therapy to the liver (e.g., ablation or embolization) within 28 days prior to randomization.
3. ECOG performance status > 2 (see Appendix IV).
4. Non-healing wound, skin ulcers, or incompletely healed bone fracture.
5. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to planned start of study therapy.
6. History of bleeding from esophageal and/or gastric varices or high risk of bleeding from varices seen on endoscopy (normal EGD required within 6 months of randomization).
7. History of GI perforation, abdominal fistulae, or intra-abdominal abscess.
8. Significant cardiovascular disease:

   1. New York Heart Association cardiac disease (Class II or greater),
   2. Myocardial infarction, unstable angina or cerebrovascular accident within past 3 months,
   3. Unstable arrhythmia,
   4. Poorly controlled arterial hypertension (defined as systolic blood pressure (BP) > 150 mmHg and/or diastolic blood pressure > 100 mmHg) based on an average of > 3 BP readings on > 2 sessions), or prior history of hypertensive crisis or hypertensive encephalopathy,
   5. Aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis within 6 months prior to randomization
9. Known contraindication to Bevacizumab or Immune Checkpoint Inhibitor (ICI): Active or history of autoimmune disease or immune deficiency, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, autoimmune hypophysitis, or autoimmune pancreatitis. Includes known hypersensitivity to any component of Bevacizumab; Chinese hamster ovary cell products or other recombinant human or humanized antibodies. Known hypersensitivity to Atezolizumab or any of the excipients. (Note: Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone and those with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study).
10. Known history of (Human immunodeficiency virus (HIV), HBV and HCV co-infection). For patients with active HBV: HBV DNA <500IU/mL obtained within 28 days prior to randomization and anti-HBV treatment (per local standard of care, e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study.
11. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
12. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis.
13. Active tuberculosis.
14. Prior allogeneic stem cell or solid organ transplantation.
15. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
16. Recent administration of live vaccine.
17. History of malignancy other than HCC within 5 years prior to screening, with the exception of adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ of breast, or Stage I uterine cancer.
18. Treatment with strong CYP3A4 inducers within 14 days prior to randomization.
19. Treatment with an immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 14 days prior to randomization, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: a) patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy), or b) patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency.
20. Current or recent (within 7 days of randomization) use of aspirin (325mg/day), dipyramidole, ticlopidine, clopidogrel, or cilostazol, Vitamin K antagonists, direct oral anticoagulants (DOACs), LMWH.
21. Recent history (within 4 weeks) of hemoptysis.
22. History of TIA, CVA, or any arterial thrombotic event within 12 months before randomization.
23. Sensory/motor neuropathy greater than or equal to grade 2, as defined by the NCI CTCAE and history of hypomagnesemia.
24. Known severe allergic reaction to contrast (e.g., anaphylaxis).
25. Pregnancy or lactating women.
26. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Hepatectomy | 17 Weeks
  Proportion of patients who undergo hepatectomy in each arm (number of patients who undergo hepatectomy divided by the number of patients randomized to each arm).

SECONDARY OUTCOMES:
Response rate | 2 years
  Radiological and pathological response rate to neoadjuvant therapy.
Toxicity to SBRT | 2 years
  Toxicity rate related to neoadjuvant SBRT.
Postoperative complications | 90 days post operatively
  Postoperative complication rate and mortality
Survival Progression Free | 2 years
  Progression free survival (PFS).
Survival | 2 years
  Overall survival (OS).
Toxicity to Atezolizumab/Bevacizumab | 2 years
  Toxicity to Atezolizumab/Bevacizumab in the neoadjuvant setting

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Meyers, MD, Principal Investigator — principle investigator; Jim Wright, MD, Study Director — OCOG Director
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - 8. Centre the recherche du Centre hospitalier de l'Université de Montréal - CHUM, Montreal, Quebec
  - McGill Cedars Cancer Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No